CLINICAL TRIAL: NCT02037425
Title: Exploratory Study of the Natural History, Clinical Outcomes, and Neuronal Endplate Changes in Subjects Reporting Short Duration vs. Long Duration of Benefit for OnabotulinumtoxinA in Treatment of Chronic Migraine
Brief Title: Duration of Benefit for OnabotulinumtoxinA in Treatment of Chronic Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cady, Roger, M.D. (Individual)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-002AL
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Results first posted 2016-03-08 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Migraine
Keywords: Chronic Migraine; onabotulinumtoxinA; Headache; Migraine; Neuronal regrowth; Botox
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- onabotulinumtoxinA (Other): At visit 2, subjects will receive their first treatment at Day 29 (+/-3 days). All subjects will receive 155 U Botulinum Toxin Type A Purified Neurotoxin Complex administered at 31 fixed-site, fixed-dose injections across seven (7) specific head/neck muscle areas. Injections will be repeated at day 113 (+/- 3 days) and at day 197 (+/- 3 days).
  Interventions: Drug: onabotulinumtoxinA

INTERVENTIONS:
Drug: onabotulinumtoxinA — BOTOX® (Formulation Number 9060X) contains 200 International Units (IU) of Clostridium botulinum Toxin Type A, reconstituted with 4 cc of normal saline providing 5 units per 0.1 cc. At visit 2, subjects will receive their first treatment at Day 29 (+/-3 days). All subjects will receive 155 U Botulinum Toxin Type A Purified Neurotoxin Complex administered at 31 fixed-site, fixed-dose injections across seven (7) specific head/neck muscle areas. Injections will be repeated at day 113 (+/- 3 days) and at day 197 (+/- 3 days).
  Other Names: Botox

SUMMARY:
To obtain a patient specific understanding of response to treatment with onabotulinumtoxinA by collecting and correlating pre and post treatment subject specific history, clinical outcomes, and histological changes.

DETAILED DESCRIPTION:
Recognizing a commitment to evidence-based science as the pathway to optimize clinical outcomes for patients with chronic migraine (CM) we believe this investigator initiated study (IIS) will:

1. Help clinicians recognize the importance of scheduling patients with CM at intervals not exceeding 12 weeks.
2. Provide biopsy evidence supporting sensory mechanisms involved in the mechanism of action (MOA) of onabotulinumtoxinA (BTX). This does not exclude potential valuable contributions of denervation of motor neurons, but may support a more balanced and understandable mechanism for BTX in treating CM.
3. Provide clinicians important educational information for patients to better manage expectations of using BTX in managing CM and answering critical questions such as:

   1. How long does it take for BTX to begin providing a clinical benefit?
   2. What is the expected duration of this benefit?

      * Failure to understand unmet expectations either real or otherwise results in defining BTX treatment as a failure by patients and/or clinicians.
4. Provide validation for patients' reports of shorter duration of action of BTX so patients will not be misinterpreted as non-responders to BTX prematurely.
5. Ascertain if subjects initially reporting short duration of BTX response continue to experience this similar pattern of effect with repeated injection cycles.
6. Provide the first detailed longitudinal assessment of BTX response.
7. Correlate the onset and duration of benefit for subjects receiving BTX.
8. Observe factors predictive of duration of BTX response.

This study proposes to accomplish these goals through an exploratory comparison of the clinical efficacy and natural history of BTX measured at weekly time intervals. Subjects reporting short (<10 weeks) duration of benefit and subjects reporting long (>10 weeks) duration of clinical benefit will provide the primary comparison. Histological examinations (in a subset of subjects) of neuronal changes associated with regeneration of terminal neuronal endplates will be used to support these clinical observations. This study will follow subjects through 3 injection cycles or 36 weeks. Biopsies will be performed on consenting subjects prior to their first and second injection cycles.

Group Assignment

At Visit 3, subjects will be assigned to one of three groups (Groups A, B, C) based on their answers to the following questions:

1. Since your last BTX treatment, do you think there has been improvement in your chronic migraine? If the answer to Q1 is yes, subject will answer Q2 and Q3. If the answer is no, subject is assigned to Group C and no further answers are required:
2. How many days did it take for you to first notice benefit from BTX injections?
3. How long did you feel you received benefit from BTX (number of weeks)?

Subjects will be assigned into 3 groups:

1. Group A are subjects reporting 10 or less weeks of benefit from BTX;
2. Group B are subjects reporting >10 weeks of benefit from BTX;
3. Group C are subjects reporting no or minimal (< 30%) benefit from BTX.

Consistency of subjects' perception of BTX benefit at 12 weeks will be compared to responses at 24 and 36 weeks, though Group assignment will remain as defined at 12 weeks.

This exploratory study will be conducted at the Headache Care Center in Springfield, MO. Thirty-six subjects, 18 years and older with a history of chronic migraine will be enrolled. The study will consist of 5 visits for all subjects.

At Visit 1 (day 1 of baseline) the following study procedures will be performed:

* Informed Consent obtained
* Migraine, medical and medication history obtained
* Physical and neurological exam performed
* Urine pregnancy test performed if applicable
* Vital signs collected

At Visit 2 (day 29 +/- 3 days) the following study procedures will be performed:

* Update medical and medication history
* Urine pregnancy test performed if applicable
* Vital signs collected
* Review baseline diary
* Complete Migraine Disability Assessment Scale (MIDAS)
* Complete Social Readjustment Rating Scale (SRRS)
* Complete Beck Depression Inventory II (BDI-II)
* Complete State-Trait Anxiety Inventory (STAI)
* Complete Sleep Quality Questionnaire
* Punch biopsy for neuronal regrowth (subset of subjects)
* onabotulinumtoxinA injections

At Visit 3 (day 113 +/- 3 days) the following study procedures will be performed:

* Update medical and medication history
* Urine pregnancy test performed if applicable
* Vital signs collected
* Complete Subject Global Impression of Change (SGIC)
* Complete Physician Global Impression of Change (PGIC)
* Complete Migraine Disability Assessment Scale (MIDAS)
* Complete Social Readjustment Rating Scale (SRRS)
* Complete Beck Depression Inventory II (BDI-II)
* Complete State-Trait Anxiety Inventory (STAI)
* Complete Sleep Quality Questionnaire
* Complete duration of response to onabotulinumtoxinA questions
* Punch biopsy for neuronal regrowth (subset of subjects)
* onabotulinumtoxinA injections

At Visit 4 (day 197 +/- 3 days) the following study procedures will be performed:

* Update medical and medication history
* Urine pregnancy test performed if applicable
* Vital signs collected
* Complete Subject Global Impression of Change (SGIC)
* Complete Physician Global Impression of Change (PGIC)
* Complete Migraine Disability Assessment Scale (MIDAS)
* Complete Social Readjustment Rating Scale (SRRS)
* Complete Beck Depression Inventory II (BDI-II)
* Complete State-Trait Anxiety Inventory (STAI)
* Complete Sleep Quality Questionnaire
* Complete duration of response to onabotulinumtoxinA questions
* onabotulinumtoxinA injections

At Visit 5 (day 281 +/- 3 days) the following study procedures will be performed:

* Update medical and medication history
* Urine pregnancy test performed if applicable
* Vital signs collected
* Complete Subject Global Impression of Change (SGIC)
* Complete Physician Global Impression of Change (PGIC)
* Complete Migraine Disability Assessment Scale (MIDAS)
* Complete Social Readjustment Rating Scale (SRRS)
* Complete Beck Depression Inventory II (BDI-II)
* Complete State-Trait Anxiety Inventory (STAI)
* Complete Sleep Quality Questionnaire
* Complete duration of response to onabotulinumtoxinA questions

ELIGIBILITY:
Inclusion Criteria:

* male or female 18 years or older.
* able to read, understand, and sign the informed consent.
* a negative urine pregnancy test at visit 1, if female, and of childbearing potential. Note: If female of childbearing potential, subject must agree to maintain true abstinence or use one of the listed methods of birth control for the duration of the study: hormonal contraceptive, intrauterine device (IUD), condoms, diaphragm, and/or have a male partner who has undergone a successful vasectomy. The use of barrier contraceptive (condom or diaphragm) should always be supplemented with the use of a spermicide.

Note: To be considered not of childbearing potential, subject must be 6 weeks post-surgical bilateral oophorectomy, hysterectomy, bilateral tubal ligation, postmenopausal for at least one year.

* at least a one year history of migraine
* history of chronic migraine (with or without aura) according to the criteria of the International Classification of Headache Disorders (ICHD)-3 for at least 3 months prior to enrollment (Appendix I)
* able to differentiate migraine headache from any other headache they may experience (e.g., cluster headache)
* onset of migraine before age 50
* willing to provide responses to questionnaires and complete the online diary.
* if taking migraine preventive(s), be on a stable dose of the preventive medication for at least 30 days prior to screening
* concomitant medication dosages approved by the investigator
* email and internet access for completion of online diary

Exclusion Criteria:

* previously used onabotulinumtoxinA as a migraine preventative or has used onabotulinumtoxinA for any other reason during the prior year
* female who is pregnant, planning to become pregnant during the study period, breast feeding, or is of childbearing potential and not practicing a reliable form of birth control
* headache disorders outside ICHD-3 defined chronic migraine that cannot be easily distinguished from CM (Appendix I)
* evidence of underlying pathology contributing to their headaches
* any medical condition that may increase their risk with exposure to BTX including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other significant disease that might interfere with neuromuscular function
* profound atrophy or weakness of muscles in the target areas of injection
* skin conditions or infections at any of the injection sites
* allergy or sensitivities to any component of the test medication
* in the opinion of the investigator, has an active major psychiatric disorder including substance abuse and/or substance dependence within the last 12 months as determined by the investigator.
* Medication Overuse Headache as defined by ICHD-3 criteria for opioid or butalbital containing products (Appendix II)
* planning or requiring surgery during the study
* a history of poor compliance with medical treatment
* currently participating in an investigational drug study or has participated in an investigational drug study within the previous 30 days of the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger K Cady, M.D., Principal Investigator — Clinvest
Locations (1):
- Clinvest/A Division of Banyan Group, Inc., Springfield, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | onabotulinumtoxinA
Started | 44
Randomized to Treatment | 32
Completed | 18
Not Completed | 26

BASELINE CHARACTERISTICS:
Population: 44 subjects screened, 3 subjects failed inclusion/exclusion at screening, 9 subjects did not meet criteria after baseline. 32 subjects randomized to treatment. While 32 subjects randomized and were used for reporting demographics, two subjects didn't complete any outcome measures, therefore only 30 participants were used for endpoint analysis.
Groups:
- onabotulinumtoxinA: At visit 2, subjects will receive their first treatment at Day 29 (+/-3 days). All subjects will receive 155 U Botulinum Toxin Type A Purified Neurotoxin Complex administered at 31 fixed-site, fixed-dose injections across seven (7) specific head/neck muscle areas. Injections will be repeated at day 113 (+/- 3 days) and at day 197 (+/- 3 days). A total of 30 subjects were used in data analysis as 2 subjects did not complete any outcome measures once enrolled in the study.
Arm/Group | onabotulinumtoxinA
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.56 (9.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Subject Global Impression of Change
Description: Changes in the Subject's Global Impression of Change (SGIC) measured at weeks 12, 24, and 36 for Groups A, B, and C. Subject global impression of change was measured on a 7 point scale with 0 being Very Much Worse and 7 Very Much Improved.
Time Frame: Weeks 12, 24, and 36 Post Randomization
Population: Subjects included in this outcome measure analysis include those completing treatment period 1 injection cycle and returning at visit 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group A: Subjects reporting 10 weeks or less of benefit from onabotuliunumtoxinA.
- Group B: Subjects reporting greater than 10 weeks of benefit from onabotuliunumtoxinA.
- Group C: Subjects reporting no or minimal of benefit from onabotuliunumtoxinA (3 weeks or less).
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 21 | 3 | 6
units on a scale
  Week 12 Post Randomization | 4.43 (1.94) | 5.67 (0.47) | 1.67 (1.80)
  Week 24 Post Randomization | 4.76 (1.38) | 5.33 (0.47) | 3.33 (1.60)
  Week 36 Post Randomization | 4.14 (2.17) | 5.33 (0.47) | 2.50 (1.80)

2. Primary Outcome: Duration of onabotulinumtoxinA Over 3 Injection Cycles in Groups A, B, and C
Description: Compare the duration of onabotulinumtoxinA response through the 3 injection cycles of the study for Groups A, B, and C as measured by headache days during each period (Baseline (28 days), Treatment Period 1(84 days), Treatment Period 2(84 days), and Treatment Period 3(84 days). Duration of response is defined as a 30% reduction in the number of headache days compared to baseline.
Time Frame: From day 29 (first day of injection cycle 1) to day 281 (84th day of injection cycle 3) plus or minus 12 days
Measure: Number; unit: percentage of responders
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 21 | 3 | 6
percentage of responders
  Treatment Period 1 | 62 | 67 | 0
  Treatment Period 2 | 62 | 100 | 50
  Treatment Period 3 | 62 | 100 | 50

3. Secondary Outcome: Headache Days
Description: Comparison of headache days per month over each injection cycle between Groups A, B, and C (Baseline (28 days), Treatment Period 1(84 days), Treatment Period 2(84 days), and Treatment Period 3(84 days). Subjects will remain in their assigned groups based on assessment at 12 weeks.
Time Frame: From day 29 (first day of injection cycle 1) to day 281 (84th day of injection cycle 3) plus or minus 12 days
Measure: Mean (Standard Deviation); unit: number of headache days
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 21 | 3 | 6
number of headache days
  Baseline | 21.95 (4.19) | 22.33 (2.36) | 24.83 (3.02)
  Treatment Period 1 | 44.76 (19.80) | 37.0 (10.61) | 64.83 (11.71)
  Treatment Period 2 | 35.06 (21.27) | 29.33 (12.66) | 55 (21.88)
  Treatment Period 3 | 31.43 (22.0) | 29.33 (12.66) | 65.67 (22.43)

4. Secondary Outcome: Migraine Disability Assessment Scale (MIDAS)
Description: Comparison between Group A, B, and C for MIDAS total scores (effect migraine headaches have on subjects daily function) measured at baseline and weeks 12, 24, and 36.
  Total score of disability ranges:
  * 0 to 5, MIDAS Grade I, Little or no disability
  * 6 to 10, MIDAS Grade II, Mild disability
  * 11 to 20, MIDAS Grade III, Moderate disability
  * 21+, MIDAS Grade IV, Severe disability Score ranges from 0-450. No subscales are present.
Time Frame: Baseline, Week 12, Week 24, and Week 36 Post Randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 21 | 3 | 6
units on a scale
  Baseline | 84.19 (54.60) | 115.67 (55.26) | 74.33 (56.78)
  Week 12 Post Randomization | 19.90 (14.44) | 25.67 (11.12) | 96.83 (70.07)
  Week 24 Post Randomization | 27.65 (22.03) | 28.00 (5.89) | 66.33 (44.54)
  Week 36 Post Randomization | 28.29 (28.35) | 30.33 (15.80) | 86.00 (40.56)

5. Secondary Outcome: Social Readjustment Rating Scale (SRRS)
Description: Comparison between Group A, B, and C for SRRS scores (impact of common stressors) measured at baseline and weeks 12, 24, and 36. Scores can range from 0 to an undetermined amount, as subjects are allowed to rate unlisted events according to their own sense of stress. A total lower than 150 suggests a low level of stress and a low probability of developing a stress-related disorder. Scores greater than 150 suggest higher levels of stress and higher probabilities of developing stress-related disorders.
Time Frame: Baseline, Week 12, Week 24, and Week 36 Post Randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 21 | 3 | 6
units on a scale
  Baseline | 168.68 (108.77) | 157.00 (81.86) | 199.50 (161.30)
  Week 12 Post Randomization | 131.76 (115.98) | 168.33 (57.05) | 141.67 (99.60)
  Week 24 Post Randomization | 85.33 (81.33) | 215.33 (163.94) | 122.50 (138.08)
  Week 36 Post Randomization | 81.81 (93.02) | 221.00 (117.29) | 70.83 (87.49)

6. Secondary Outcome: Physician Global Impression of Change (PGIC)
Description: Comparison between Group A, B, and C for PGIC scores measured at weeks 12, 24, and 36. the PGIC scale scores range from 0-7 with 0 being Very Much Worse and 7 being Very Much Improved. A higher score indicates a greater impression of change.
Time Frame: Week 12, Week 24, and Week 36 Post Randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 21 | 3 | 6
units on a scale
  Week 12 Post Randomization | 4.95 (1.05) | 5.33 (0.47) | 3.50 (1.26)
  Week 24 Post Randomization | 5.00 (1.02) | 5.33 (0.47) | 4.00 (0.58)
  Week 36 Post Randomization | 4.81 (1.10) | 5.00 (0.82) | 3.67 (0.94)

7. Secondary Outcome: Beck Depression Inventory II (BDI-II)
Description: Comparison between Group A, B, and C for BDI-II scores measured at baseline and weeks 12, 24, and 36. A total score of 0-10 = these ups and downs are considered normal, 11-16 = mild mood disturbance,17-20 = borderline clinical depression, 21-30 = moderate depression, 31-40 = severe depression, over 40 = extreme depression
Time Frame: Baseline, Week 12, Week 24, and Week 36 Post Randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 21 | 3 | 6
units on a scale
  Baseline | 11.62 (10.27) | 16.67 (6.13) | 11.83 (6.41)
  Week 12 Post Randomization | 8.43 (9.20) | 11.00 (3.27) | 7.67 (2.92)
  Week 24 Post Randomization | 7.48 (9.10) | 12.33 (5.44) | 7.00 (4.97)
  Week 36 Post Randomization | 9.00 (9.19) | 7.00 (4.97) | 7.00 (4.04)

8. Secondary Outcome: State-Trait Anxiety Inventory (STAI)
Description: Comparison between Group A, B, and C for STAI scores measured at baseline and weeks 12, 24, and 36. Scores range from 20-80, with 20 indicating lower levels of anxiety most generally, and 80 indicating higher levels of anxiety most generally.
Time Frame: Baseline, Week 12, Week 24, and Week 36 Post Randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 21 | 3 | 6
units on a scale
  Baseline | 38.76 (17.97) | 43.67 (13.89) | 40.67 (7.25)
  Week 12 Post Randomization | 36.05 (10.08) | 40.00 (6.53) | 36.50 (8.64)
  Week 24 Post Randomization | 36.62 (9.73) | 38.00 (11.43) | 38.00 (6.16)
  Week 36 Post Randomization | 36.86 (9.92) | 36.33 (6.94) | 38.33 (8.79)

9. Secondary Outcome: Sleep Quality Question
Description: Comparison between Group A, B, and C for sleep quality scores measured at baseline and weeks 12, 24, and 36 post-randomization. A single sleep quality question was asked indicating quality of sleep over the past four weeks. The scale ranged from 1-5, with 1 being very poor quality and 5 being very good quality of sleep.
Time Frame: Baseline, Week 12, Week 24, and Week 36 Post Randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 21 | 3 | 6
units on a scale
  Baseline | 3.19 (1.01) | 3.33 (0.47) | 3.00 (0.58)
  Week 12 Post Randomization | 3.48 (0.85) | 3.67 (0.47) | 2.5 (0.50)
  Week 24 Post Randomization | 3.57 (0.95) | 3.33 (0.47) | 2.83 (0.69)
  Week 36 Post Randomization | 3.38 (1.05) | 3.67 (1.25) | 2.50 (0.76)

10. Secondary Outcome: Acute Medication Usage
Description: Comparison of acute medication usage between Groups A, B, and C during baseline, Treatment Period 1, 2, and 3.
Time Frame: From day 1 (first day of baseline) to day 281 (84th day of injection cycle 3) plus or minus 12 days
Measure: Mean (Standard Deviation); unit: number of medications used
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 21 | 3 | 6
number of medications used
  Baseline | 16.29 (10.92) | 12.00 (5.10) | 13.83 (5.46)
  Treatment Period 1 | 36.53 (24.26) | 20.67 (9.03) | 36.00 (19.72)
  Treatment Period 2 | 28.33 (20.98) | 26.33 (10.08) | 28.33 (16.02)
  Treatment Period 3 | 25.71 (18.77) | 9.67 (6.60) | 28.00 (16.39)

11. Secondary Outcome: Consistency of Response to onbotulinumtoxinA Over Three Injection Cycles
Description: Compare the consistency of duration of onabotulinumtoxinA response by the group assignment at 12 weeks to assessments at 24, and 36 weeks evaluations as measured by the number of responders. A responder is defined as a 30% reduction from baseline in the number of headache days.
Time Frame: Weeks 12, 24, and 36 Post Randomization
Measure: Number; unit: participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 21 | 3 | 6
participants
  Treatment Period 1 | 13 | 2 | 0
  Treatment Period 2 | 13 | 3 | 3
  Treatment Period 3 | 13 | 3 | 3

12. Secondary Outcome: Duration of onabotulinumtoxinA Over 3 Injection Cycles
Description: Compare duration of benefit of onabotulinumtoxinA response through 3 injection cycles as measured by headache days per week (including the last 4 weeks of every injection cycle). A percent of responders was calculated using a 30% reduction of the number of headache days compared to average number of headache per week during baseline.
Time Frame: Weeks 9, 10, 11, 12, 21, 22, 23, 24, 33, 34, 35, 36 Post Randomization
Measure: Number; unit: percentage of responders
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 21 | 3 | 6
percentage of responders
  Week 9 Post Randomization | 57 | 33 | 33
  Week 10 Post Randomization | 57 | 67 | 17
  Week 11 Post Randomization | 52 | 67 | 0
  Week 12 Post Randomization | 38 | 67 | 17
  Week 21 Post Randomization | 76 | 67 | 33
  Week 22 Post Randomization | 62 | 67 | 50
  Week 23 Post Randomization | 57 | 100 | 50
  Week 24 Post Randomization | 52 | 67 | 33
  Week 33 Post Randomization | 62 | 67 | 33
  Week 34 Post Randomization | 71 | 100 | 33
  Week 35 Post Randomization | 48 | 100 | 33
  Week 36 Post Randomization | 48 | 100 | 17

13. Other Pre Specified Outcome: Neuronal Regrowth
Description: Compare neuronal regrowth in the skin biopsies with duration of benefit of onabotulinumtoxinA in Groups A, B, C from baseline to 12 weeks post randomization. Neuronal regrowth change was scored on a 0-3 point scale with 0 being no change from baseline in regrowth and 3 being significant change from baseline.
Time Frame: Baseline & Week 12 Post Randomization
Population: Only a subset of subjects (n = 14) completed this endpoint for the trial based on the protocol design.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 9 | 2 | 3
units on a scale
  Beta Tublin | .61 (.66) | 0.0 (0.0) | 1.17 (1.02)
  Calcitonin Gene-Related Peptide | 1.06 (1.01) | 0.0 (0.0) | 1.0 (1.41)
  SNAP25 (Synaptosomal-Associated Protein) | 1.22 (1.03) | 0.5 (0.5) | 0.67 (0.47)

ADVERSE EVENTS:
Time Frame: From day 1 (first day of baseline) to day 281 (84th day of injection cycle 3) plus or minus 12 days
Arm/Group | onabotulinumtoxinA
Serious Adverse Events (participants affected / at risk) | 2/44
Other Adverse Events (participants affected / at risk) | 23/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | onabotulinumtoxinA (N=44)
Dizziness (Nervous system disorders) | 1 (1)
Expressive Aphasia (Nervous system disorders) | 1 (1)
Unsteady Gait (Nervous system disorders) | 1 (1)
Spontaneous Abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | onabotulinumtoxinA (N=44)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Eyebrow Droop (Musculoskeletal and connective tissue disorders) | 3 (3)
Eyebrow Heaviness (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Sinus Infection (Infections and infestations) | 2 (2)
Strep Throat (Infections and infestations) | 4 (4)
Upper Respiratory Infection (Infections and infestations) | 3 (3)
Weight Gain (Metabolism and nutrition disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes